CLINICAL TRIAL: NCT00095043
Title: A 12-Month, Randomized, Double-Blind, Placebo-Controlled, Parallel Groups, Multicenter Long-Term Safety Study of MK0928 in the Treatment of Elderly Outpatients With Primary Insomnia
Brief Title: Safety of MK0928 on Insomnia in the Elderly (0928-005)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0928-005; MK0928-005; 2004_088
Record Dates: First submitted 2004-10-29; First posted 2004-11-01 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — gaboxadol

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0928, gaboxadol
Drug: Comparator: placebo

SUMMARY:
The purpose of this trial is to study the safety of MK0928 on insomnia in the elderly.

DETAILED DESCRIPTION:
The duration of treatment is 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Insomnia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 320
Dates: Start 2004-10; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability after 12 months of treatment

SECONDARY OUTCOMES:
Discontinuation symptoms and rebound insomnia using sleep diary and Tyrer Withdrawal Symptom Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC